CLINICAL TRIAL: NCT04521530
Title: A Comparative Study Between Immediate Functional and Non-functional Loading of Dental Implants in the Posterior Alveolar Mandibular Region (a Randomized Clinical Trial)
Brief Title: Immediate Functional Versus Non Functional Implant Loading in the Mandible
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant lecturer, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Dental implants
Record Dates: First submitted 2020-08-18; First posted 2020-08-20 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Dental Implants; Edentulous Alveolar Ridge

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- immediate functional loading with temporary crowns (Experimental): patients were rehabilitated with immediate functionally loaded implants.
  Interventions: Other: immediate functional implant loading
- immediate non functional loading with temporary crowns (Experimental): patients were rehabilitated with immediate non-functionally loaded implants.
  Interventions: Other: immediate non functional implant loading

INTERVENTIONS:
Other: immediate functional implant loading — Patients will undergo implant placement and a minimum of 35 Ncm reading with the graded torque wrench. Temporary crowns in functional occlusion were cemented.
  Arms: immediate functional loading with temporary crowns
Other: immediate non functional implant loading — implant will be placed into the site following the manufacturer's protocol making sure to have a minimum of 35 Newton centimeter reading with the degraded torque wrench. Non-functional temporary crowns were cemented.
  Arms: immediate non functional loading with temporary crowns

SUMMARY:
comparing immediate functionally loaded implants and immediate non functionally loaded implants in the posterior mandibular region on bases of bone density and bone loss evaluated by cone-beam computed tomography (CBCT).

DETAILED DESCRIPTION:
Patients are more demanding after the revolution in immediate implant dentistry which reduces implant procedure nowadays according to literature and research. In response to patients' demands not only implants are immediately placed but also immediately loaded within 72 hours reducing the time for prosthetic loading and also improving bone formation according to some studies. The debate in modern implant dentistry is whether to immediately load the implants in functional occlusion or non-functional occlusion and which will improve the osseointegration and reduce crestal bone loss.

Implants of the BioInfinity system were placed in 16 subjects divided into two groups.

Group (A): 8 patients with missing posterior mandibular teeth whom will be rehabilitated with immediate functionally loaded implants.

Group (B): 8 patients with missing posterior mandibular teeth in whom immediate non-functionally loaded implants were used.

The two groups were evaluated at baseline, immediately after implant placement and 4 months postoperative to evaluate crestal bone level and quantitative radiographic bone density using CBCT.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged (20-40) years old.
* Missing Posterior tooth or teeth indicated for implant placement.
* Residual alveolar ridge at least 10 mm high and at least 4 mm wide.

Exclusion Criteria:

* Systemic diseases that will contraindicate the surgery.
* Poor Oral Hygiene.
* The patient refuses to undergo the surgery.
* Parafunctional habits.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-29 (Actual)

PRIMARY OUTCOMES:
Pain score | immediately Postoperatively
  Visual analogue scale consist of a scale of 10 0 means no pain 10 menas pain is as bad as it could possibly be
Change in crestal bone loss | immediately Postoperatively and after 4 months
  CBCT was done immediately after implant placement and 4 months postoperatively to assess crestal bone loss

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt